CLINICAL TRIAL: NCT05091697
Title: Cost-utility of the Multicomponent Program VIRTUAL FIBROWALK in Patients With Fibromyalgia
Brief Title: Cost-utility of VIRTUAL FIBROWALK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Universitat Autonoma de Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COST-UTILITY VIIRTUAL FW
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Fibromyoma;Cervix
Keywords: Cost-utility; Fibromyalgia; multicomponent treatment; randomized controlled trial
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent treatment VIRTUAL FIBROWALK + TAU (Experimental): VIRTUAL FIBROWALK is a multicomponent non-pharmacological program based on Pain Neuroscience Education (PNE), therapeutic exercise, Cognitive Behavioural Therapy (CBT) and Mindfulness Training
  Interventions: Behavioral: Multicomponent treatment VIRTUAL FIBROWALK + TAU
- Treatment as Usual (TAU) (Active Comparator): Treatment-as-Usual (TAU) consisted of the prescribed drugs adapted to the symptomatic profile of each patient and basic face to face and written advice on PNE and aerobic exercise adapted to the physical capacities of the patients at the beginning of the study.patient
  Interventions: Behavioral: Multicomponent treatment VIRTUAL FIBROWALK + TAU

INTERVENTIONS:
Behavioral: Multicomponent treatment VIRTUAL FIBROWALK + TAU — To assess the effectiveness and cost-utility of the virtual multicomponent program (Fibrowalk)

SUMMARY:
The main objective of this study is to assess the effectiveness and cost-utility of the VIRTUAL FIBROWALK multicomponent treatment program as coadjuvant of treatment-as- usual (TAU) compared to TAU alone.

DETAILED DESCRIPTION:
This is a two-arm RCT focused on the effectiveness and cost-utility of the multicomponent program VIRTUAL FIBROWALK as coadjuvant of treatment-as- usual (TAU) vs. TAU alone (in a 3-month follow-up RCT) VIRTUAL FIBROWALK combines multicomponent approach based on Pain Neuroscience Education (PNE), therapeutic exercise, Cognitive Behavioural Therapy (CBT) and Mindfulness training.

ELIGIBILITY:
Inclusion Criteria:

* Adults from 18 to 75 years-old.
* 1990 American College of Rheumatology (ACR) classification criteria + the 2011 modified ACR diagnostic criteria for fibromyalgia
* Able to understand Spanish and accept to participate in the study.

Exclusion Criteria:

* Participating in concurrent or past RCTs (previous year).
* Comorbidity with severe mental disorders (i.e. psychosis) or neurodegenerative diseases (i.e. Alzheimer) that that would limit the ability of the patient to participate in the RCT.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2021-12-10 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Revised Fibromyalgia Impact Questionnaire (FIQR) | Change from baseline values at 6 months
  The FIQR comprises three dimensions: physical dysfunction (scores from 0 to 30), overall impact (scores from 0 to 20), and intensity of the symptoms (scores from 0 to 50) is used to measure the impact generated by FM during the last week. It consists of 21 items, which are answered on a numerical rating scale of 11 points (from 0 to 10). Total scores can range from 0 to 100, with higher scores reflecting greater deterioration.
Client Service Receipt Inventory (CSRI) | Change from baseline values at 6 months
  The Client Service Receipt Inventory (CSRI) is a tool used to collect information on the whole range of services and supports study participants may use. This data can be used for a wide range of applications, including estimating the costs of service receipt.
EuroQoL questionnaire (EQ-5D-5L) | Change from baseline values at 6 months
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.

SECONDARY OUTCOMES:
Tampa Scale for Kinesiophobia (TSK-11) | Change from baseline values at 6 months
  TSK-11 is used to assess fear of pain and movement. It consists of 11 items, which are answered on a Likert scale of 4 points. Total scores of each scale range from 11 to 44, where higher scores indicate a greater fear of pain and movement.
Hospital Anxiety and Depression Scale (HADS) | Change from baseline values at 6 months
  HADS is used to quantify the severity of anxiety and depression symptoms. It consists of two dimensions (anxiety and depression) of 7 items each responding on a Likert scale of 4 points. Total scores of each scale (HADS-A and HADSD) range from 0 to 21, where higher scores indicate greater severity of symptoms.
Physical Function of the 36-Item Short Form Survey (SF-36) | Change from baseline values at 6 months
  Physical Function of the 36-Item Short Form Survey (SF-36) was used to measure physical function.This dimension comprises a total of 10 items, which are answered on a Likert scale of 3 points. Total scores on each scale are then transformed and can range from 0 to 100, with higher scores indicate better physical function.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayte Serrat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No